CLINICAL TRIAL: NCT00615030
Title: A Phase III Randomized, Double Blind, Double Dummy, Placebo Controlled, Multicenter, 4 Treatments, 3 Period Incomplete Block Crossover Study to Assess the Efficacy and Safety of Indacaterol 300 µg o.d. Dosed in the Evening in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD), Using Salmeterol 50 µg b.i.d. as Active Control
Brief Title: Study of Indacaterol Dosed in the Evening in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2305
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, bronchodilator, long acting beta agonist, LABA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (12):
- Indacaterol Morning,Indacaterol Evening, Salmeterol (Experimental): In period I, indacaterol 300 μg once a day in the morning delivered via single dose dry powder inhaler (SDDPI) with a placebo to salmeterol delivered via dry powder inhaler (DPI). Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period II, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period III, Salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and second dose in the evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol Evening,Indacaterol Morning, Placebo (Experimental): In period I, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period II, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period III, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Salmeterol, Placebo, Indacaterol Morning (Experimental): In period I, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose was in the evening along with placebo matching indacaterol delivered by SDDPI. In period II, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period III, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Placebo, Salmeterol, Indacaterol Evening (Experimental): In period I, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period II, salmeterol 50 μg twice daily delivered via dry powder inhaler (DPI). One of the two daily doses of salmeterol was administered in the morning and the second dose was in the evening along with placebo matching indacaterol delivered by SDDPI. In period III, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via dry DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol Morning, Placebo, Indacaterol Evening (Experimental): In period I, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period II, During morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period III, Patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol Evening,Salmeterol, Indacaterol Morning (Experimental): In period I, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period II, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period III, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Salmeterol, Indacaterol Evening, Placebo (Experimental): In period I, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period II, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period III, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Placebo, Indacaterol Morning, Salmeterol (Experimental): In period I, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period II, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via dry powder inhaler DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period III, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol Morning, Salmeterol, Placebo (Experimental): In period I, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period II, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period III, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Indacaterol Evening, Placebo, Salmeterol (Experimental): In period I, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via dry powder inhaler DPI. In period II, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period III, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Salmeterol, Indacaterol Morning, Indacaterol Evening (Experimental): In period I, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period II, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period III, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol
- Placebo, Indacaterol Evening, Indacaterol Morning (Experimental): In period, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period II, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period III, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol

INTERVENTIONS:
Drug: Indacaterol — 300 µg dosed in the morning/evening via single dose dry powder inhaler (SDDPI)
  Other Names: QAB149
Drug: Salmeterol — 50 µg twice daily delivered via dry powder inhaler (DPI)
  Other Names: Serevent®
  Arms: Indacaterol Evening, Placebo, Salmeterol; Indacaterol Evening,Salmeterol, Indacaterol Morning; Indacaterol Morning, Salmeterol, Placebo; Indacaterol Morning,Indacaterol Evening, Salmeterol; Placebo, Indacaterol Morning, Salmeterol; Placebo, Salmeterol, Indacaterol Evening; Salmeterol, Indacaterol Evening, Placebo; Salmeterol, Indacaterol Morning, Indacaterol Evening; Salmeterol, Placebo, Indacaterol Morning
Drug: Placebo to Indacaterol — Placebo matching indacaterol was delivered via SDDPI.
Drug: Placebo to Salmeterol — Placebo matching salmeterol was delivered via DPI

SUMMARY:
This study was conducted to provide detailed information on the efficacy of indacaterol (in terms of the spirometry assessment forced expiratory volume in 1 second [FEV1]) over the full 24-h time period

ELIGIBILITY:
Inclusion criteria:

* Male and female adults aged ≥ 40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure
* Co-operative outpatients with a diagnosis of chronic obstructive pulmonary disease (COPD) (moderate to severe as classified by the Global initiative for chronic obstructive lung disease (GOLD) Guidelines, 2006) and:
* Smoking history of at least 20 pack years
* Post-bronchodilator FEV1 < 80% and ≥30% of the predicted normal value
* Post-bronchodilator FEV1/forced vital capacity (FVC) < 70%

Exclusion criteria:

* Pregnant or lactating females
* Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to Visit 1 or during the run-in period
* Patients requiring long term oxygen therapy (>15 h a day)
* Patient who have had a respiratory tract infection 6 weeks prior to V2 (with further criteria)
* Patients with concomitant pulmonary disease, pulmonary tuberculosis, or clinically significant bronchiectasis
* Patients with history of asthma (with further criteria)
* Patients with Type I or uncontrolled type II diabetes.
* Patients who have clinically relevant laboratory abnormalities or a clinically significant abnormality
* Any patient with active cancer or a history of cancer with less than 5 years disease free survival time
* Patient with a history with long QT syndrome or whose QTc interval is prolonged
* Patients with a hypersensitivity to any of the study drugs or drugs with similar chemical structure
* Patients who have had treatment with an investigational drug (with further criteria)
* Patients who have had live attenuated vaccination within 30 days prior to Visit 2, or during run-in period
* Patients with known history of non compliance to medication
* Patients unable to satisfactorily use a dry powder inhaler device or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — + 41 61 324 1111
Locations (7):
- France (2):
  - Novartis Investigative Site, Beuvry
  - Novartis Investigative Site, Nantes
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Barcelona, Spain

REFERENCES:
- [Derived] Magnussen H, Verkindre C, Jack D, Jadayel D, Henley M, Woessner R, Higgins M, Kramer B; INPUT study investigators. Indacaterol once-daily is equally effective dosed in the evening or morning in COPD. Respir Med. 2010 Dec;104(12):1869-76. doi: 10.1016/j.rmed.2010.08.010. Epub 2010 Sep 20. PMID 20850959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to one of the 12 possible treatment sequences of the double-blind 10-week treatment phase (Week 1 - 10). Each treatment sequence was divided into three treatment periods (I/II/III) of 15-day duration each. The first and second treatment period of each sequence was followed by a 2-week washout period.
Pre-assignment Details: Total 96 patients were randomized; one randomized patient discontinued from the study prior to exposure to study drug because of abnormal test procedure(s) result.
Groups:
- Sequence 1:Indacaterol Morning,Indacaterol Evening, Salmeterol: In period I, indacaterol 300 μg once a day in the morning delivered via single dose dry powder inhaler (SDDPI) with a placebo to salmeterol delivered via dry powder inhaler (DPI). Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period II, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period III, Salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and second dose in the evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 2:Indacaterol Evening,Indacaterol Morning, Placebo: In period I, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period II, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period III, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 3: Salmeterol, Placebo, Indacaterol Morning: In period I, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose was in the evening along with placebo matching indacaterol delivered by SDDPI. In period II, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period III, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 4: Placebo, Salmeterol, Indacaterol Evening: In period I, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period II, salmeterol 50 μg twice daily delivered via dry powder inhaler (DPI). One of the two daily doses of salmeterol was administered in the morning and the second dose was in the evening along with placebo matching indacaterol delivered by SDDPI. In period III, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via dry DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 5: Indacaterol Morning, Placebo, Indacaterol Evening: In period I, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period II, During morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period III, Patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 6:Indacaterol Evening,Salmeterol, Indacaterol Morning: In period I, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period II, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period III, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 7: Salmeterol, Indacaterol Evening, Placebo: In period I, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period II, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period III, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 8: Placebo, Indacaterol Morning, Salmeterol: In period I, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period II, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via dry powder inhaler DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period III, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 9:Indacaterol Morning, Salmeterol, Placebo: In period I, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period II, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period III, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 10: Indacaterol Evening, Placebo, Salmeterol: In period I, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period II, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period III, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 11:Salmeterol,Indacaterol Morning,Indacaterol Evening: In period I, salmeterol 50 μg twice daily delivered via DPI. One of the two daily doses of salmeterol was administered in the morning and the second dose in evening along with placebo matching indacaterol delivered by SDDPI. In period II, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. In period III, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Sequence 12: Placebo, Indacaterol Evening, Indacaterol Morning: In period, during morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. In period II, patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via SDDPI with placebo to salmeterol delivered via DPI. In period III, indacaterol 300 μg once a day in the morning delivered via SDDPI with a placebo to salmeterol delivered via DPI. Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
Period: Period I
Arm/Group | Sequence 1:Indacaterol Morning,Indacaterol Evening, Salmeterol | Sequence 2:Indacaterol Evening,Indacaterol Morning, Placebo | Sequence 3: Salmeterol, Placebo, Indacaterol Morning | Sequence 4: Placebo, Salmeterol, Indacaterol Evening | Sequence 5: Indacaterol Morning, Placebo, Indacaterol Evening | Sequence 6:Indacaterol Evening,Salmeterol, Indacaterol Morning | Sequence 7: Salmeterol, Indacaterol Evening, Placebo | Sequence 8: Placebo, Indacaterol Morning, Salmeterol | Sequence 9:Indacaterol Morning, Salmeterol, Placebo | Sequence 10: Indacaterol Evening, Placebo, Salmeterol | Sequence 11:Salmeterol,Indacaterol Morning,Indacaterol Evening | Sequence 12: Placebo, Indacaterol Evening, Indacaterol Morning
Started | 9 | 8 | 9 | 8 | 9 | 6 (1 randomized patient in this sequence dropped out before exposure to study drug in Period I.) | 7 | 7 | 9 | 8 | 8 | 7
Completed | 8 | 8 | 9 | 8 | 8 | 5 | 7 | 7 | 8 | 8 | 7 | 6
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Administrative problem | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Abnormal laboratory value(s) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period II
Arm/Group | Sequence 1:Indacaterol Morning,Indacaterol Evening, Salmeterol | Sequence 2:Indacaterol Evening,Indacaterol Morning, Placebo | Sequence 3: Salmeterol, Placebo, Indacaterol Morning | Sequence 4: Placebo, Salmeterol, Indacaterol Evening | Sequence 5: Indacaterol Morning, Placebo, Indacaterol Evening | Sequence 6:Indacaterol Evening,Salmeterol, Indacaterol Morning | Sequence 7: Salmeterol, Indacaterol Evening, Placebo | Sequence 8: Placebo, Indacaterol Morning, Salmeterol | Sequence 9:Indacaterol Morning, Salmeterol, Placebo | Sequence 10: Indacaterol Evening, Placebo, Salmeterol | Sequence 11:Salmeterol,Indacaterol Morning,Indacaterol Evening | Sequence 12: Placebo, Indacaterol Evening, Indacaterol Morning
Started | 8 | 8 | 9 | 8 | 8 | 5 | 7 | 7 | 8 | 8 | 7 | 6
Completed | 8 | 8 | 8 | 7 | 8 | 5 | 6 | 7 | 7 | 8 | 7 | 6
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject withdrew consent | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | Sequence 1:Indacaterol Morning,Indacaterol Evening, Salmeterol | Sequence 2:Indacaterol Evening,Indacaterol Morning, Placebo | Sequence 3: Salmeterol, Placebo, Indacaterol Morning | Sequence 4: Placebo, Salmeterol, Indacaterol Evening | Sequence 5: Indacaterol Morning, Placebo, Indacaterol Evening | Sequence 6:Indacaterol Evening,Salmeterol, Indacaterol Morning | Sequence 7: Salmeterol, Indacaterol Evening, Placebo | Sequence 8: Placebo, Indacaterol Morning, Salmeterol | Sequence 9:Indacaterol Morning, Salmeterol, Placebo | Sequence 10: Indacaterol Evening, Placebo, Salmeterol | Sequence 11:Salmeterol,Indacaterol Morning,Indacaterol Evening | Sequence 12: Placebo, Indacaterol Evening, Indacaterol Morning
Started | 8 | 8 | 8 | 7 | 8 | 5 | 6 | 7 | 7 | 8 | 7 | 6
Completed | 7 | 8 | 8 | 6 | 8 | 5 | 6 | 7 | 7 | 8 | 7 | 6
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative problems | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Patients
Number analyzed (Participants) | 95
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures were based on safety population.
  years | 64.1 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 80

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) Following 14 Days of Evening Dosing of Indacaterol Versus Placebo
Description: Trough FEV1 was assessed by performing spirometry measurements in the clinic for each treatment period. For the primary efficacy variable, trough FEV1 is the mean of two measurements taken at 23h 10 min and 23h 45 min post dose. The primary variable was analyzed using an analysis of covariance (ANCOVA) model with the (period) baseline FEV1 as covariate.
  The (period) baseline FEV1 was defined as the value measured before the study drug administration in that treatment period.
Time Frame: After 14 days of treatment
Population: The modified intention-to-treat (mITT) population included all randomized patients who received at least one dose of study drug. Patients who received only one treatment were also included for calculation of treatment means. This analysis included all patients who received indacaterol in the evening or placebo in their assigned treatment sequence.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol Evening: Patients were instructed to take morning doses of a placebo to indacaterol delivered via single dose dry powder inhaler (SDDPI) and placebo to salmeterol delivered via dry powder inhaler (DPI). Indacaterol 300 μg once a day in the evening delivered via single dose dry powder inhaler (SDDPI) with placebo to salmeterol delivered via dry powder inhaler (DPI). Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Placebo: During evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
Arm/Group | Indacaterol Evening | Placebo
Number analyzed (Participants) | 63 | 64
Liters | 1.57 (0.025) | 1.37 (0.025)

2. Secondary Outcome: Trough FEV1 Assessed After 14 Days of Dosing for All Other Treatment Comparisons
Description: Trough FEV1 was assessed by performing spirometry measurements in the clinic for each treatment period. On the morning and evening of Day 15 trough FEV1 (i.e. mean of measurements performed 23 h 10 min and 23 h 45 min post-dose) were assessed. An analysis of covariance (ANCOVA) model was used with the (period) baseline FEV1 as covariate. The (period) baseline FEV1 was defined as the value measured before the study drug administration in that treatment period.
Time Frame: After 14 days of dosing
Population: The modified intention-to-treat (mITT) population included all randomized patients who received at least one dose of study drug. Patients who received only one treatment were also included for calculation of treatment means.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol Morning: Indacaterol 300 μg once a day in the morning delivered via single dose dry powder inhaler (SDDPI) with a placebo to salmeterol delivered via dry powder inhaler (DPI). Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Indacaterol Evening: Patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via single dose dry powder inhaler (SDDPI) with placebo to salmeterol delivered via dry powder inhaler (DPI). Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Salmeterol Morning: In the morning, Salmeterol 50 μg delivered via dry powder inhaler (DPI) along with placebo matching indacaterol via SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Salmeterol Evening: In the evening, Salmeterol 50 μg delivered via dry powder inhaler (DPI) along with placebo matching indacaterol via SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Placebo Morning; Placebo Evening: Placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via manufacturer's proprietary DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
Arm/Group | Indacaterol Morning | Indacaterol Evening | Salmeterol Morning | Salmeterol Evening | Placebo Morning | Placebo Evening
Number analyzed (Participants) | 65 | 63 | 65 | 65 | 66 | 64
Liters | 1.56 (0.025) | 1.57 (0.025) | 1.51 (0.025) | 1.46 (0.025) | 1.36 (0.025) | 1.37 (0.025)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: In the safety population, all patients were analyzed according to treatment received.
Groups:
- Indacaterol Evening: Patients were instructed to take morning doses of a placebo to indacaterol delivered via SDDPI and placebo to salmeterol delivered via DPI. Indacaterol 300 μg once a day in the evening delivered via single dose dry powder inhaler (SDDPI) with placebo to salmeterol delivered via dry powder inhaler (DPI). Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. All patients were provided with a SABA for use (if needed) as rescue medication throughout the study.
- Indacaterol Morning: Indacaterol 300 μg once a day in the morning delivered via single dose dry powder inhaler (SDDPI) with a placebo to salmeterol delivered via dry powder inhaler (DPI). Patients were also instructed to take evening doses of a placebo to indacaterol via SDDPI and placebo to salmeterol via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. All patients were provided with a SABA for use (if needed) as rescue medication throughout the study.
- Salmeterol: Salmeterol 50 μg twice daily delivered via dry powder inhaler (DPI). One of the two daily doses of salmeterol was administered in the morning along with placebo matching indacaterol delivered by single dose dry powder inhaler (SDDPI). The second dose of salmeterol was administered in the evening along with placebo matching indacaterol delivered by SDDPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. All patients were provided with a SABA for use (if needed) as rescue medication throughout the study.
- Placebo: During morning and evening, placebo matching indacaterol was delivered via SDDPI and placebo matching salmeterol was delivered via DPI. Daily inhaled corticosteroid treatment (if applicable) was allowed to remain stable throughout the study. All patients were provided with a SABA for use (if needed) as rescue medication throughout the study.
Arm/Group | Indacaterol Evening | Indacaterol Morning | Salmeterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/65 | 1/68 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 10/65 | 4/68 | 3/68 | 5/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Evening (N=65) | Indacaterol Morning (N=68) | Salmeterol (N=68) | Placebo (N=68)
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Evening (N=65) | Indacaterol Morning (N=68) | Salmeterol (N=68) | Placebo (N=68)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.